CLINICAL TRIAL: NCT01804569
Title: The Effects of Self-Moxibustion Therapy on Subjective Physical Symptoms and Health-related Quality of Life of the Elderly.
Brief Title: The Effects of Self-Moxibustion Therapy on Subjective Physical Symptoms and Health-related Quality of Life of the Elderly. The Effects of Self-Moxibustion Therapy
Acronym: moxa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University (Other)
Responsible Party: Principal Investigator, Jooshin Kim, PhD candidate, Pusan National University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: moxa201097603
Record Dates: First submitted 2013-03-02; First posted 2013-03-05 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: Health Improvement of the Elderly
MeSH Terms: interventions — Moxibustion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- moxa (Experimental): moxibustion treatment 3 times a week for 3 weeks
  Interventions: Other: moxibustion

INTERVENTIONS:
Other: moxibustion — modernly developed moxibustion treatment device with safe cover on top of it.
  Other Names: Shinkigoo (신기구); company: bosungsa

SUMMARY:
There will be significant differences between control and experimental group after the moxibustion intervention as to, subjective physical symptoms and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Male and female older adults age between 65-85
* Agree to participate and sign for the trail after understanding of study purpose, and method.
* Able to answer for questions by verbally or literally
* Able to participate in 2weeks after follow-up

Exclusion Criteria:

* Having physical disorder such as thyroids, severe heart disease, dietetic mellitus, severe liver disease, allergy
* Subjects who can not attend more than 3 times of intervention session
* Subjects who are eligible by the decision of investigator

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
subjective physiological symptoms | 2 weeks after the intervention

SECONDARY OUTCOMES:
Quality of Life | 2 weeks after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jooshin Kim, MSW, Principal Investigator — Pusan National University